CLINICAL TRIAL: NCT01785810
Title: A Phase II Study to Assess the Efficacy of Maraviroc in Prophylaxis of GVHD in Patients With Hematologic Malignancies Undergoing Reduced-Intensity Allogeneic SCT From Unrelated Donors
Brief Title: Phase II Maraviroc for GVHD Prevention
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UPCC 04712
Record Dates: First submitted 2013-02-05; First posted 2013-02-07 (Estimated); Results first posted 2021-01-11 (Actual); Last update posted 2021-01-11 (Actual); Status verified 2020-12

CONDITIONS: Hematologic Malignancy
MeSH Terms: conditions — Hematologic Neoplasms | interventions — Maraviroc

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Maraviroc (Experimental): Phase II, single arm, single center trial, assessing the efficacy of the combination of tacrolimus, methotrexate and maraviroc as graft-versus-host disease (GVHD) prophylaxis after unrelated donor peripheral blood stem-cell transplantation in patients with hematologic malignancies. Patients enrolled on this trial will receive a standard conditioning regimen with fludarabine and busulfan followed by a peripheral blood stem cell infusion from an unrelated donor, standard GVHD prophylaxis and standard antiviral and antifungal prophylaxis. In addition, all patients will receive maraviroc from day -3 to d+ 90.
  Interventions: Drug: Maraviroc 300 mg

INTERVENTIONS:
Drug: Maraviroc 300 mg — Patients enrolled on this trial will receive a standard conditioning regimen with fludarabine and busulfan followed by a peripheral blood stem cell infusion from an unrelated donor, standard GVHD prophylaxis and standard antiviral and antifungal prophylaxis. In addition, all patients will receive maraviroc from day -3 to d+ 90.
  Other Names: CCR5 Antagonist

SUMMARY:
RATIONALE: Successful allogeneic stem-cell transplantation is often limited by graft-versus-host disease (GVHD). Migration of donor cells into tissues plays a major role in GVHD. Drugs that block chemokine receptors such as CCR5, can potentially decrease the migration of donor cells into tissues. Blocking CCR5 after allogeneic stem-cell transplantation may therefore reduce the rates of GVHD.

PURPOSE: This study explores the efficacy of pharmacologic inhibition of CCR5 in prevention of GVHDby administering maraviroc during allogeneic stem-cell transplantation with reduced intensity conditioning.

DETAILED DESCRIPTION:
Detailed Description:

PRIMARY OBJECTIVES:

To estimate the cumulative incidence of grade 2-4 acute GVHD by day 180 with the addition of maraviroc to a standard prophylaxis regimen in patients with hematologic malignancies undergoing reduced intensity allogeneic stem-cell transplantation (RIC SCT) from unrelated donors.

SECONDARY OBJECTIVES:

1. To assess the toxicity of a prolonged administration of maraviroc in patients undergoing RIC SCT.
2. To estimate the rates of severe (grade 3-4) acute GVHD by day 100 and 180, grade 2-4 acute GVHD by day 100, organ-specific acute GVHD, chronic GVHD, relapse, infections, non-relapse mortality, use of immunosuppressive therapies and 1-year survival in patients treated with maraviroc after RIC SCT.
3. To assess the effect of treatment with maraviroc on immune recovery, engraftment and donor T-cell chimerism in peripheral blood and in target organs.
4. To assess the effect of donor and recipient CCR5 genotype on the incidence of acute GVHD in patients receiving maraviroc as part of a GVHD prophylaxis regimen.

OUTLINE: Patients receive a standard conditioning regimen with fludarabine and busulfan followed by a peripheral blood stem cell infusion from an unrelated donor, standard GVHD prophylaxis and standard antiviral and antifungal prophylaxis. In addition, all patients receive maraviroc from day -3 to d+ 90.

Patients are followed for 1 year after the stem-cell infusion.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥18 years of age with a hematologic malignancy other than aplastic anemia or primary myelofibrosis, scheduled to undergo RIC allogeneic SCT with a peripheral blood stem cell graft from an unrelated donor, using Flu/Bu conditioning and Tac/MTX GVHD prophylaxis. The following diagnoses are included:

  * Acute leukemia - AML, ALL or acute biphenotypic leukemia. Patients will have documentation of complete remission within 6 weeks prior to their transplant. Complete remission is defined as <5% blasts on a bone marrow biopsy and absence of any known extramedullary disease.
  * Chronic myelogenous leukemia in any stage, but with documentation of <5% blasts on a bone marrow biopsy within 6 weeks prior to transplant.
  * Myelodysplastic syndrome of any subtype, but with documentation of <5% blasts on a bone marrow biopsy within 6 weeks prior to transplant.
  * Myeloproliferative disorders other than primary myelofibrosis.
  * Lymphoma - All types of lymphoma are eligible.
  * CLL and PLL.
* Patients who meet institutional eligibility criteria for allogeneic SCT:

  * Renal function: Serum creatinine ≤2.
  * Hepatic function: Baseline direct bilirubin, ALT or AST lower than three times the upper limit of normal.
  * Pulmonary disease: FVC or FEV1 ≥ 40% predicted.
  * Cardiac ejection fraction ≥ 40%.
* Availability of an unrelated donor, identified and screened by the NMDP. The donor will have at least 7/8 HLA-A, -B, -C and -DRB1 matching by high resolution molecular typing and will meet NMDP eligibility criteria to serve as a peripheral blood stem-cell donor.
* Karnofsky score ≥ 70% at the time of screening.
* Capacity to understand and sign the study informed consent form.
* Negative pregnancy test. Women of childbearing potential (not having had a hysterectomy, a bilateral oophorectomy or bilateral tubal ligation, or be post-menopausal with a total cessation of menses of > 1 year) must agree to use documented reliable method(s) of contraception. Men should agree to use condoms during the study period.

  * Co-enrollment in other clinical trials that do not include experimental GVHD therapies is allowed.

Exclusion Criteria

* Patients with aplastic anemia or primary myelofibrosis. Patients with marrow fibrosis secondary to MDS, AML or a myeloproliferative disorder other than primary myelofibrosis are eligible.
* Patients who are not expected to be available for follow-up in our institution for at least 180 days after the transplant.
* Prior allogeneic SCT.
* Uncontrolled bacterial, viral or fungal infections.
* Patients who receive maraviroc for the treatment of HIV infection.
* Patients receiving other investigational drugs for GVHD.
* Co-enrollment in other clinical trials that do not include experimental GVHD therapies is allowed.
* Patients with prior malignancies are excluded unless treated with curative intent and known to be free of disease for at least 2 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2013-02 (Actual); Primary Completion 2016-11-11 (Actual); Study Completion 2018-07-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Porter, MD, Principal Investigator — Abramson Cancer Center at Penn Medicine
Locations (1):
- Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Maraviroc: Maraviroc - 300 mg
Period: Overall Study
Arm/Group | Maraviroc
Started | 37
Completed | 29
Not Completed | 8

BASELINE CHARACTERISTICS:
Groups:
- Maraviroc: Maraviroc 300 mg
Arm/Group | Maraviroc
Number analyzed (Participants) | 37
Age, Continuous [Mean (Full Range); unit: years] | 65 [49 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 23
Comorbidity Index [Count of Participants; unit: Participants] — The comorbidity index indicates the presence of other medical conditions that increase the risk of hospitalization or death. The high category indicates a score >2.
  Participants
    Low | 7
    Intermediate | 12
    High | 18
Diagnosis [Count of Participants; unit: Participants]
  Acute myeloid leukemia | 27
  Myelodysplastic syndrome | 6
  Non-Hodgkin's lymphoma | 1
  Myeloproliferative neoplasms | 1
  Acute lymphoblastic leukemia | 2
Donor [Count of Participants; unit: Participants]
  Matched unrelated | 31
  Single-antigen mismatched | 6
Donor Age [Mean (Full Range); unit: years] | 32 [19 to 53]
Cytomegalovirus Serostatus [Count of Participants; unit: Participants]
  Recipient positive | 18
  Donor positive | 9
  Negative | 10
CD34+ cell dose [Mean (Full Range); unit: x 10^6 cells/kg] | 6.2 [1.5 to 20.2]
Disease Risk Index [Count of Participants; unit: Participants] — The disease risk index uses information about the underlying disease and disease status to categorize patients according to risk of relapse and survival.
  Participants
    Low | 3
    Intermediate | 16
    High/very high | 18
Donor Sex [Count of Participants; unit: Participants]
  Male | 24
  Female | 13
CD3+ cell dose [Mean (Full Range); unit: x 10^8 cells/kg] | 2.2 [0.6 to 8.1]
CD4+ cell dose [Mean (Full Range); unit: x 10^8 T cells/kg] | 1.5 [0.3 to 5.4]
CD8+ cell dose [Mean (Full Range); unit: x 10^8 T cells/kg] | 0.7 [0.1 to 2.2]

OUTCOME MEASURES:

1. Primary Outcome: Day +180 Rate of Grade II-IV Acute GVHD
Description: The cumulative incidence of grade II-IV acute GVHD by day 180 after the stem-cell infusion. This is based on consensus conference criteria.
Time Frame: 180 days
Measure: Count of Participants; unit: Participants
Arm/Group | Maraviroc
Number analyzed (Participants) | 37
Participants | 22

ADVERSE EVENTS:
Time Frame: From the initiation of maraviroc (Day -3) to d+ 120 days following stem-cell infusion.
Groups:
- Maraviroc: Maraviroc - dose level of 300 mg
Arm/Group | Maraviroc
Serious Adverse Events (participants affected / at risk) | 5/37
Other Adverse Events (participants affected / at risk) | 29/37
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Maraviroc (N=37)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pericardial effusion (Cardiac disorders) | 1 (1)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 2 (2)
Sepsis (Infections and infestations) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Maraviroc (N=37)
Anemia (Blood and lymphatic system disorders) | 7
Febrile Neutropenia (Blood and lymphatic system disorders) | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 5
Pericardial effusion (Cardiac disorders) | 1
Diarrhea (Gastrointestinal disorders) | 4
Esophagitis (Gastrointestinal disorders) | 1
Dysgeusia (Nervous system disorders) | 1
Hypoglycemia (Metabolism and nutrition disorders) | 1
Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 3
Oral pain (Gastrointestinal disorders) | 1
Rectal mucositis (Gastrointestinal disorders) | 1
White blood cell decreased (Investigations) | 7
Hypomagnesemia (Metabolism and nutrition disorders) | 3
Hypokalemia (Metabolism and nutrition disorders) | 2
Aspartate aminotransferase increased (Investigations) | 3
Prolonged partial thromboplastin time (Investigations) | 4
Hypocalcemia (Metabolism and nutrition disorders) | 4
Nausea (Gastrointestinal disorders) | 4
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2
Anorexia (Metabolism and nutrition disorders) | 4
Dehydration (Metabolism and nutrition disorders) | 3
Hyperkalemia (Metabolism and nutrition disorders) | 3
Hypophosphatemia (Metabolism and nutrition disorders) | 2
Fatigue (General disorders) | 4
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1
Lymphocyte count decreased (Investigations) | 7
Peripheral sensory neuropathy (Nervous system disorders) | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 2
Alanine aminotransferase increased (Investigations) | 3
Hypercalcemia (Investigations) | 1
INR Increased (Investigations) | 3
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2
Hyperbilirubinemia (Investigations) | 3
Edema limbs (General disorders) | 2
Hypotension (Vascular disorders) | 2
Oral mucositis (Gastrointestinal disorders) | 5
Constipation (Gastrointestinal disorders) | 2
Hemorrhoids (Gastrointestinal disorders) | 1
Headache (Nervous system disorders) | 1
Depression (Psychiatric disorders) | 1
Dizziness (Nervous system disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 6
Alkaline phosphatase increased (Investigations) | 1
Decreased platelets (Investigations) | 7
Rectal pain (Gastrointestinal disorders) | 1
Dysphagia (Gastrointestinal disorders) | 1
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Creatinine Elevated (Investigations) | 4
Sore throat (Respiratory, thoracic and mediastinal disorders) | 2
Hematuria (Renal and urinary disorders) | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 3
Neutropenia (Investigations) | 7
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Multi-organ failure (General disorders) | 1
Anxiety (Psychiatric disorders) | 2
Fever (General disorders) | 1
Bladder spasm (Renal and urinary disorders) | 1
Flushing (Vascular disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Bloating (Gastrointestinal disorders) | 1
Abdominal distension (Gastrointestinal disorders) | 1
Tumor lysis syndrome (Metabolism and nutrition disorders) | 1
Depressed level of consciousness (Nervous system disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Urinary retention (Renal and urinary disorders) | 1
Hypermagnesemia (Metabolism and nutrition disorders) | 1
Flatulence (Gastrointestinal disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Rash maculopapular (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No